CLINICAL TRIAL: NCT00183911
Title: Phase II Study of Adjuvant Intraperitoneal FUDR Treatment Added to Chemoradiation (5-Fluorouracil/Leucovorin Plus Total Dose 4500 cGy of External Beam Radiotherapy) in Patients With Fully Resected Locally Advanced Gastric Adenocarcinoma
Brief Title: Study of 5-Fluorouracil and Leucovorin and Intra-abdominal Floxuridine Chemoradiation in Patients With Fully Resected Locally Advanced Gastric Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH); New York University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3G-03-1
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Gastric Adenocarcinoma; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Floxuridine; Fluorouracil; Leucovorin; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: floxuridine, 5-Fluorouracil, leucovorin
Procedure: External Beam Radiotherapy
Procedure: Surgery

SUMMARY:
The purpose of this study is to evaluate the side effects of a new treatment for stomach cancer which may potentially improve the prognosis of this cancer.

Our principle objective is to improve the results of standard chemotherapy and radiation after surgery of patients with gastric cancer. The intra-abdominal (intraperitoneal) administration of floxuridine (FUDR) is a procedure that we have studied and have determined it is a safe treatment. In this study, we want to evaluate the side effects of this treatment when it is given after surgery but before standard intravenous chemotherapy and radiation.

Study treatment will start with surgical removal of the part of the stomach with cancer, together with surrounding tissues and lymph nodes. After surgery, patients will get treatment with a chemotherapy drug, FUDR, administered directly into the abdomen. This is called intraperitoneal chemotherapy. After this treatment patients will receive repeated intravenous injection of two drugs, 5-fluorouracil and leucovorin alone or combined with irradiation of the abdomen.

ELIGIBILITY:
Inclusion Criteria:

* Histologic dx of locally advanced gastric adenocarcinoma (requires upper endoscopy with bx of lesion and CT scan of chest, abdomen, and pelvis with iv and oral contrast or other methods of imaging to confirm absence of metastatic dz) (Untreated patients with histologically documented gastric/GEJ ca stages IB-IV [M0] are eligible)
* Based on post-op pathological findings, diagnosis and staging has to confirm stage IB-IV (M0) adenocarcinoma of stomach or GEJ.
* Patients who underwent emergency surgery for indications such as GI obstruction, perforation, or hemorrhage, or patients with surgery already performed, are eligible provided surgery is considered curative
* ECOG performance status 0-2
* AGC greater than or equal to 1.5; platelets greater than or equal to 100,000; Hgb greater than or equal to 9.0· Total bilirubin less than or eqal to 2.0; SGOT/SGPT less than or equal to 2.5 x uln; alk phos less than or equal to 2.5 x uln
* BUN less than or equal to 30; creatinine less than or equal to 1.5 or CrCl >60 ml/min
* Negative b-HCG pregnancy test (females with reproductive potential)
* PT, aPTT, and thrombin time within range of normal
* Evidence of at least unilateral renal function as established by CT scan with contrast or nephrogram. (If only one kidney is present, at least 2/3 of the functioning kidney must be excluded from any RT port)

Exclusion Criteria:

* Prior radiation therapy, chemotherapy or immunotherapy
* Presence of another active invasive malignancy (Except for adequately treated basal cell or squamous cell skin ca, in-situ cervical ca, or other cancer for which patient has been disease-free for at least 5 yrs)
* Active or uncontrolled infection, including HIV
* Psychiatric disorders that would interfere with informed consent· Pregnant or nursing women (Patients of reproductive age must agree to use effective contraceptive method)
* Any other severe concurrent disease, which in the judgment of MD would make patient inappropriate for study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2003-11; Primary Completion 2006-12 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Syma Iqbal, M.D., Study Chair — U.S.C./Norris Comprehensive Cancer Center
Locations (1):
- U.S.C. / Norris Comprehensive Cancer Center, Los Angeles, California, United States